CLINICAL TRIAL: NCT04095806
Title: Zanzibar Stroke Study. Using a Prospective Register-based Study, Qualitative Research, and Economic Analysis to Support Evidence Synthesis for Health Policy and System Change in Zanzibar, Tanzania.
Brief Title: Zanzibar Stroke Study: Narrowing the Gaps in Hypertension Care, and Improving Stroke Outcomes (ZanStroke)
Acronym: ZanStroke
Status: Completed | Type: Observational
Sponsor: Jutta Mari Adelin Jorgensen (Other)
Collaborators: Newcastle University, UK (Unknown); Vervig (IoM) (Unknown)
Responsible Party: Sponsor-Investigator, Jutta Mari Adelin Jorgensen, Principal Investigator of ZanStroke, Dr. Jutta Mari Adelin Jorgensen, Mnazi Mmoja National Referral Hospital
Organization: Mnazi Mmoja National Referral Hospital (Other)
Other Study IDs: ZAHREC/02/July/2019/47
Record Dates: First submitted 2019-09-18; First posted 2019-09-19 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample separated into fractions (RBC, buffy coat, plasma), serum, and whole blood will be stored for future studies (not part of the ZanStroke study)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Stroke (exposure) — stroke case definition (exposure) listed in inclusion/exclusion criteria section

SUMMARY:
Background:

A previous study in Zanzibar (which Jutta Adelin Jorgensen, PI of ZanStroke, led) showed a high prevalence of hypertension among adults at 33%, in fact higher than average in Sub-Saharan Africa (SSA), and poor performance of the health systems with nearly 90% of people with hypertension not achieving adequate blood pressure control. Uncontrolled hypertension (HTN) and stroke have already become among the commonest causes of admission to and death at hospital in Zanzibar. At the same time, there is little or no data available to quantify the stroke burden on types, treatment and outcomes, cost of stroke care, nor a comprehensive understanding of the causes of poor hypertension control in the population.The Tanzanian Stroke Incidence study (which Richard Walker from Newcastle University led) showed some of the highest stroke incidence rates in the world. However, there are many unanswered questions, and the Zanzibar Stroke Study will be a unique opportunity to look at all stroke admissions from a large island population.

Zanzibar Stroke Study:

The hypotheses investigated are

1a. Current challenges in stroke care cannot exclusively be explained by limited structural resources, and care delivering processes play an essential role.

1. b. Current organization and quality of care for stroke including rehabilitation could benefit from being aligned with best practices for low resource settings.
2. a. Stroke types, causes, and prognosis are dominated by a higher proportion of hemorrhagic strokes, associated to poorly controlled hypertension, higher 30-day mortality, and worse prognosis in terms of disability and mortality at 12 months than seen in high income settings.

2b Long term stroke outcome is not only depending on stroke severity but also on sociodemographic/economic factors with worse prognosis for the poorest part of the population.

3a. There is a significant first stage delay due to local perceptions and beliefs around stroke which prohibits biomedical treatment in the prognostically important acute phase of stroke 3b. There are untapped resources in the community that could be leveraged to increase adherence to medical treatment to control BP to prevent stroke and re-stroke, as well as making rehabilitation accessible 4a. Introducing a hypertension care package at lowest primary care level for people at high cardiovascular disease (CVD) risk to prevent stroke and re-stroke is cost-effective, affordable, and possible.

4b. With no intervention, the cost of stroke care at hospital level will in 10 years exceed the cost of all reproductive and child health (RCH) services.

ZanStroke is an observational, prospective study of stroke admissions to hospitals in Zanzibar (Unguja) enrolling all patients with a recent stroke (< 30 days) over a period of one year to investigate the burden of stroke disease, risk factors and outcome up till 12 months post-stroke. This will be done through establishing a stroke patient register.

Participant data will include sociodemographic and -economic information, vascular risk factors and previous medical history, routine head-CT, routine biochemical results and other investigations, as well as early and long-term outcomes (deaths, disability, independence/functionality, quality of life, cognition, medicine adherence, rehabilitation therapy, re-stroke).

Approximately 80% of stroke patients in Unguja, Zanzibar who seek hospital care are admitted to the main hospital and the nearby private hospital, and these will undergo CT head scan, but this will not be possible in all of the other six hospitals. We will take blood samples and store serum and deoxyribonucleic acid (DNA) for potential future analysis from the main hospital and the nearby private hospital only.

In addition to the clinical epidemiological research, qualitative and health economic evaluation research will be undertaken to understand stroke patients and caretakers life worlds and perspectives, health care providers skills and practices, organization and processes of stroke care at hospital level, and to define a set of most cost-effective interventions to prevent and treat stroke in the particular Zanzibar context.

DETAILED DESCRIPTION:
Current and future benefits and impacts:

With the demographic transition and population ageing in SSA rates of stroke are set to continue to increase rapidly as part of the double burden of disease (still a major burden of infectious diseases, as well as an unfinished agenda of maternal and newborn health).

Previous studies have already established a global high level of hypertension in the adult population in Zanzibar, and low performance of the health system for managing this.

It is important to identify the peculiar genomic, gene-environmental and environmental risk and protective factors for stroke occurrence, pattern, type, outcome, and current incidence velocity in SSA in order to inform preventive measures especially effective and cost-effective control of raised blood pressure/hypertension; the best model for the provision of inpatient care and rehabilitation in a resource poor environment with lack of access to dedicated stroke units and limited multidisciplinary team input; and to include the particular East Africa population in existing or future international stroke collaborations to ensure that genetic variations relevant to the population there are represented.

ELIGIBILITY:
Inclusion Criteria:

* admitted with a clinical diagnosis of stroke, or developing stroke while in hospital admitted for other cause (see below for stroke case definition)
* age above 18 year
* written consent form signed by patient, or authorized representative (spouse or caretaker)
* stroke onset < 30 days when enrolled

Exclusion Criteria:

* patient or authorized representative unable to understand the information given or being interviewed.
* CT scan not suspect of stroke despite clinical suspect

Stroke case definition:

All the following stroke categories listed below that have been submitted as the most responsible diagnosis will be included in the stroke cohort. For patients developing stroke while admitted to hospital, stroke as the second diagnosis will also be included in the cohort. Patients who previously had a stroke and are being admitted due to complications, and where stroke is not the primary diagnosis during admission, will not be included in the cohort.

Definition of stroke ( ICD-10 classification code in parenthesis) that will be used in the study for inclusion in the cohort:

(a) Intracerebral hemorrhage (I61 including all sub-codes) (b) Ischemic stroke (I63 including all sub-codes, H34.1) (c) Stroke, not specified as hemorrhagic or ischemic (I64) (d) Cerebral Venous Thrombosis, non-pyogenic (I63.6) Where CTscan is not available, the clinical diagnosis of stroke will be used, and coding will be I64 (ICD-10)

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults who get admitted to hospital in Unguja (Zanzibar) due to stroke, or develop stroke while admitted to hospital.
Sampling Method: Non-Probability Sample
Enrollment: 869 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
30 day mortality | 30 days post stroke; data collected over 12 months
  Mortality rate of stroke patients 30 days post stroke
90 days mortality | 90 days post stroke; data collected over 12 months
  Mortality rate of stroke patients 90 days post stroke
12 months mortality | 12 months post stroke; data collected over 12 months
  Mortality rate of stroke patients 12 months post stroke

SECONDARY OUTCOMES:
Disability at 30 days | 30 days post stroke; data collected over 12 months
  disability of stroke patients as measured using the modified Ranking Scale (mRS) at 30 days post stroke.
  The modified Rankin Scale (mRS) assesses disability in patients who have suffered a stroke and is compared over time to check for recovery and degree of continued disability. A score of 0 is no disability, 5 is disability requiring constant care for all needs; 6 is death.
  The mRS has been used in clinical research for over 30 years and is a common standard for assessing functional outcomes in patients with stroke.
  Multiple studies have shown that the mRS correlates with physiological indicators such as stroke type, lesion size and neurological impairment as assessed by other stroke evaluation scale
Disability at 12 months | 12 months post stroke; data collected over 12 months
  disability of stroke patients as measured using modified Rankin Scale (mRS) at 12 months post stroke. The modified Rankin Scale (mRS) assesses disability in patients who have suffered a stroke and is compared over time to check for recovery and degree of continued disability. A score of 0 is no disability, 5 is disability requiring constant care for all needs; 6 is death.
  The mRS has been used in clinical research for over 30 years and is a common standard for assessing functional outcomes in patients with stroke.
  Multiple studies have shown that the mRS correlates with physiological indicators such as stroke type, lesion size and neurological impairment as assessed by other stroke evaluation scale
Cognitive impairment at 3 and 12 months | 3 and 12 months post stroke; data collected over 12 months
  Cognitive impairment of stroke patients 3 and 12 months post stroke using the Identification and Intervention for Dementia in Elderly Africans (IDEA) cognitive screening tool .
  The first 4 items involve being able to name a bridge from a description of its use, knowing the day of the week, knowing the name of the village chief/ town mayor/ city governor and naming as many animals as possible in one minute (score 2 for ≥ 8 animals, score 1 for 4-7 animals, score 0 for 0-3 animals). Item 5 is a 10-word recall test (score 1 point for each word up to a maximum of 5 points). The sixth item is designed to measure praxis and involves a matchstick design test with scores ranging from 0 (no matchsticks placed correctly), to 3 (all four matchsticks placed correctly).
  The maximum possible score is 15 and the minimum 0, with a higher score indicating better cognitive function. 7/8 is used as a cut-off for dementia, and 10/11 a cut-off for cognitive impairment
Health related Quality of Life at 3 and 12 months | 3 and 12 months post stroke; data collected over 12 months
  Quality of life among stroke patients 3 and 12 months post stroke using the 5-level EQ-5D instrument.
  The EQ-5D is a standardized non-disease specific instrument to describe and value health-related quality of life and consist of a descriptive system and a visual analogue scale (VAS).
  The descriptive system comprises of mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels. The patient indicates his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale ( 0-10), where the endpoints are labelled 'The best health you can imagine' (0) and 'The worst health you can imagine' (10).
Medicine Adherence at 3 and 12 months | 3 and 12 months post stroke; data collected over 12 months
  Medicine adherence among stroke patients 3 and 12 months post stroke using the Medicine Adherence Questionnaire (MAQ).
  MAQ is a standardized instrument to assess intentional and un-intentional non-adherence and consist of four questions with response options yes or no. No to all responses = good adherence, while one or more Yes to responses = non-adherent. Non-adherence can be identified as mainly unintentional (factor 1) or purposeful (factor 2), or mixed.
Re-stroke at 12 months | 12 months post stroke; data collected over 12 months
  proportion of stroke patients who experience a new stroke within 12 months of previous stroke

CONTACTS AND LOCATIONS:
Overall Officials: Jutta A Jorgensen, MD, Principal Investigator — Mnazi Mmoja Hospital
Locations (8):
- Tanzania (8):
  - Kivunge District Hospital, Kinyasini, Zanzibar
  - Mnazi Mmoja Hospital, Zanzibar
  - Al Rahma Hospital, Zanzibar
  - Bububu Military Hospital, Zanzibar
  - KMKM hospital Bububu, Zanzibar
  - Makunduchi District hospital, Zanzibar
  - Tasakthaa Global Hospital, Zanzibar
  - Tawakala hospital, Zanzibar

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jorgensen JA, Matuja SS. Establishing Stroke Registers in Sub-Saharan Africa: Experiences From 2 Large Referral Hospitals in Tanzania. Stroke. 2023 Sep;54(9):e417-e418. doi: 10.1161/STROKEAHA.123.043627. Epub 2023 Jul 14. No abstract available. PMID 37449421
- [Derived] Jorgensen JMA, Christensen DL, Nielsen KK, Sadiq HS, Khan MY, Jusabani AM, Walker R. Incidence and characteristics of stroke in Zanzibar-a hospital-based prospective study in a low-income island population. Front Neurol. 2022 Jul 28;13:931915. doi: 10.3389/fneur.2022.931915. eCollection 2022. PMID 35968303